CLINICAL TRIAL: NCT04553159
Title: Autologous Adipose Derived Stem Cell Transplantation in the Treatment of Keloids. A Pilot Randomized Controlled Trial
Brief Title: Autologous Adipose Derived Stem Cells Transplantation in the Treatment of Keloids.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASOREC/060/19-UG-REC-009
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Keloid; Autologus Adipose Derived Stem Cells; Feasibility; Safety
Keywords: Adipose derived stem cells; Keloids; Stromal vascular fraction
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Intervention Model Description: This is a pilot single centre randomized controlled trail with a ratio of 1:1 conducted in the Surgical out patient of Mulago Hospital Kampala
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose Derived Stem Cell(ADSC) arm (Experimental): Participants allocated to this arm will have tumescent liposuction performed on them to obtain lipoaspirate. The lipoaspirate will then be processed to obtain the stromal vascular fraction. This Adipose derived stromal vascular fraction which contains stem cells will then be infiltrated into the keloid tissue as a single dose infiltration.
  This will be harvested and infiltrated as the whole cell pellet (stromal vascular fraction) comprising of an estimate total of 9 million ADSCs (range: 8.4-9.72; SD ± 6.6).
  Interventions: Biological: Autologous adipose derived stem cells
- Triamcinolone Acetanoide (TAC) arm (Active Comparator): Participants in this arm will receive a single dose Triamcinolone acetanoide infiltration into the keloid. This will be a single dose infiltration of 40mg/cubic centimetres of keloids.
  Interventions: Biological: Autologous adipose derived stem cells

INTERVENTIONS:
Biological: Autologous adipose derived stem cells — Once consented, tumescent liposuction will be performed and 100-300ml of lipoaspirate will be collected. The harvested lipoaspirate will be processed aseptically in theatre through centrifugation at 1200g, then the sediment will be washed with Phosphate buffered saline and then incubated at 37 degrees celsius in 0.075% Collagenase type 1a for 1 hour. This will then be washed in an equal volume of 10% Fetal Bovine Serum then filtered through a 100 micrometer cell strainer. Red cells lysed using the Red cell lysis buffer will be performed followed by washing in Phosphate buffered Saline and centrifugation and the stromal vascular fraction cell pellet collected and diluted into 5ml normal saline solution for immediate infiltration. cell counts and viability using Trypan blue will be perfomed prior to the infiltration
  Other Names: Adipose derived Stromal vasular fraction infiltration

SUMMARY:
Keloids are the most common disfiguring skin disorder affecting colored population with a prevalence of upto 16%.

Autologous adipose derived stem cells have been found to have potential therapeutic benefits however limited clinical trials have compared there role to standard therapy.

This is a pilot study that is intended to evaluate the feasibility of conducting this clinical trial comparing adipose derived stromal vascular fraction to Triamcinolone in keloid treatment. The full clinical trial is already registered under the clinical trial number NCT04391621.

The objective of this Pilot is to evaluate the feasibility of conducting a full study on the same topic.

DETAILED DESCRIPTION:
Background: Keloids affect upto 16% of Africans and often demonstrate more aggressive behaviour with poor response to existing therapies.

Adipose derived stem cells have been described to have inhibitory effects on keloid growth with several invitro studies and case series reporting promising findings.

Despite this knowledge, no clinical trial has been conducted to compare the efficacy of these adipose derived stem cells to existing standard therapy. We intend to conduct a clinical trial comparing the adipose derived stem cells to the existing standard of care here in Uganda which is Triamcinolone Acetanoide a trial that is registered under the clinical trial number NCT04391621. Before scaling up this study, we intend to evaluate the feasibility to conducting a full scale study by first piloting the same trial to a smaller number of participants.

The primary objective of this study will be to describe the feasibility and safety of adipose derived stem cells in the treatment of keloids as well as to document the process of autologous adipose derived stem cells harvesting and processing. The secondary outcome will be the clinical endpoints of keloid regression and symptom relief at the end of one month.

This will be a pilot parallel and un-blinded randomised controlled trial that will be conducted at Mulago National Referral Hospital. 6 patients will be allocated randomly into either Triamcinolone group and Adipose Derived Stem cells group. Each arm will receive the respective single dose infiltration of the selected treatment.

The patients will be followed up for three months for keloid regression and symptom relief as well as development of side effects.

Utility: This pilot study is intended to evaluate the feasibility of conducting a clinical trial on the efficacy of Autologous adipose derived stem cells in the treatment of keloids

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single keloid of 1-2cm3 as these have the highest response to any treatment administered.

Exclusion Criteria:

* Previous intra-lesional steroid injection treatment in the last three months as the effects may still be ongoing Insufficient abdominal fat pad(depth) of 3cm Confirmed bleeding disorder Ongoing systemic illness Ulceration or local keloid infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | three months
  Using the Common Terminology Criteria for Adverse events (CTCAE), we shall identify any treatment associated adverse events in both treatment arms and describe the nature and grade of the adverse events.
The procedure time in hours. | three months
  We intend to evaluate the time it will take to prepare and administer the treatment in both arms.
  The intervention arm involves three steps which are liposuction, lipo-aspirate processing as well as infiltration. We intend to evaluate the time this will take and compare it to the Active control arm which consists of one step which is the infiltration. This will help answer question on feasibility of performing this procedure as a day care procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Makerere University College of Health Sciences, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
We don't intend to share individual participant data to other researchers.

REFERENCES:
- [Background] Shaffer JJ, Taylor SC, Cook-Bolden F. Keloidal scars: a review with a critical look at therapeutic options. J Am Acad Dermatol. 2002 Feb;46(2 Suppl Understanding):S63-97. doi: 10.1067/mjd.2002.120788. PMID 11807470
- [Background] Wang X, Ma Y, Gao Z, Yang J. Human adipose-derived stem cells inhibit bioactivity of keloid fibroblasts. Stem Cell Res Ther. 2018 Feb 21;9(1):40. doi: 10.1186/s13287-018-0786-4. PMID 29467010
- [Background] Lee G, Hunter-Smith DJ, Rozen WM. Autologous fat grafting in keloids and hypertrophic scars: a review. Scars Burn Heal. 2017 Apr 6;3:2059513117700157. doi: 10.1177/2059513117700157. eCollection 2017 Jan-Dec. PMID 29799555
- [Background] Ramakrishnan VM, Boyd NL. The Adipose Stromal Vascular Fraction as a Complex Cellular Source for Tissue Engineering Applications. Tissue Eng Part B Rev. 2018 Aug;24(4):289-299. doi: 10.1089/ten.TEB.2017.0061. Epub 2017 Apr 13. PMID 28316259